CLINICAL TRIAL: NCT01939847
Title: IMAGE Study: Individualized Molecular Analyses Guide Efforts in Breast Cancer - Personalized Molecular Profiling in Cancer Treatment at Johns Hopkins
Brief Title: IMAGE Study: Personalized Molecular Profiling in Cancer Treatment at Johns Hopkins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J12129; NA_00080409 (Other: JHMIRB)
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; Breast cancer; Molecular profiling; Personalized medicine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Molecular prolfiling in tissue (Experimental): Participant's tumor will be analyzed by Foundation Medicine on their FoundationOne platform - a targeted whole exome sequencing of 182 cancer related genes (3,230 exons) as well as 37 introns from 14 genes commonly rearranged or altered in cancer via next-generation sequencing technology to provide a molecular profile for a possible treatment suggestion
  Interventions: Other: Treatment suggestion
- Molecular prolfiling in blood (No Intervention): Participant's blood sample will be analyzed by Foundation Medicine on their FoundationOne platform - a targeted whole exome sequencing of 182 cancer related genes (3,230 exons) as well as 37 introns from 14 genes commonly rearranged or altered in cancer via next-generation sequencing technology; however, this is just being done to see if it is possible to generate similar results in blood samples. We do not yet know if blood sample results may be used for treatment decision (this will be tested in a future study) and results will not be given to participants; therefore, no treatment suggestion will be given.

INTERVENTIONS:
Other: Treatment suggestion — Based on any actionable findings of the molecular profiling results, the investigators will come up with a suggestion for approved treatment or for clinical trial by referencing institutional clinical trials or potentially nationwide possibilities (www.clinicaltrials.gov).
  Arms: Molecular prolfiling in tissue

SUMMARY:
This study will test the feasibility of identifying patients who could benefit from tumor molecular profiling, of analyzing the patients' tumors in a timely (28 day) fashion, and of the identification of possible actionable mutations that are not just biologically interesting but are clinically relevant. The investigators will also examine the outcome data from patients who followed the Molecular Profiling Tumor Board suggestion compared with those who did not.

When the tissue studies are done, an additional group of patients will be enrolled to test if the same is possible in blood samples.

DETAILED DESCRIPTION:
The goal of this research study is to determine if it is possible to obtain personalized genetic information from a subject's tumor to see if physicians can use that information to make a treatment suggestion. The investigators hope to identify genes important to cancer cells that could potentially identify a more educated way to recommend therapy. It is not known if our suggestion for treatment based on genetic information will be the correct treatment choice.

Subjects and their treating doctor will have a choice about what treatment they will receive and do not have to decide to be treated with the suggestion from this study. In some cases it will not be possible to make a suggestion. For example, a suggestion for treatment will not be possible if there are technical issues, if the gene sequencing process takes longer than planned, or if no genes are identified that could help identify a treatment suggestion.

The investigators also plan to collect information about the treatment subjects receive and how their cancer responds to the treatment. This may help us to understand if our personalized suggestion improves the amount of time before their disease progresses.

In addition, blood samples will be collected for research studies. These samples are being collected to learn more about breast cancer by studying cells, genes, and gene products including their patterns and changes in the blood and tissue to help to learn how cancer develops and responds to therapy.

Any man or woman being seen at Johns Hopkins for treatment of metastatic triple negative (or behaving as triple negative) breast cancer may be eligible.

Upon conclusion of the tissue studies and in order to gain experience with and assess the feasibility of receiving blood-based results using blood sampling kits, we will enroll an additional cohort of patients with recent Foundation Medicine testing for clinical purposes and collect blood samples only for research testing. The primary objectives and analysis for this new cohort will proceed similarly as the original tissue-based cohort.

ELIGIBILITY:
MOLECULAR PROFILING IN TISSUE:

Inclusion Criteria:

* Male or Female
* 18 years of age or older
* Metastatic breast cancer and treatment with prior chemotherapy (either in adjuvant, neoadjuvant or metastatic setting)
* Triple negative clinical phenotype (ER-, PR-, HER2-). For HER2 assessment, a negative result is an immunohistochemical (IHC staining of 0 or 1+, a FISH result of less than 4.0 HER2 gene copies per nucleus, or a FISH ratio of less than 1.8. ER/PR will be assessed by IHC and will be defined as positive/negative using the American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) Guidelines. Estrogen receptor (ER) and progesterone receptor (PR) assays will be considered positive if there are at least 1% positive tumor nuclei in the sample on testing in the presence of expected reactivity of internal (normal epithelial elements) and external controls. NOTE: A triple negative clinical phenotype based upon the patient's clinical course may also be eligible as determined at the discretion of the Study Chair (ie, if a patient is behaving clinically as ER/PR negative but does not meet the strict criteria outlined.)
* Patients must have a tumor suitable for biopsy and be deemed medically appropriate to undergo a biopsy
* Able to voluntarily provide informed consent

Exclusion Criteria:

* N/A

MOLECULAR PROFILING IN BLOOD:

Inclusion Criteria:

* Male or Female
* 18 years of age or older
* Metastatic breast cancer
* Any phenotype of breast cancer is eligible for enrollment (i.e., any ER, PR, and HER2 status).
* Able to voluntarily provide informed consent

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09-19 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Time to report molecular profiling in tissue | 28 days
  To demonstrate the feasibility of real-time molecular profiling of metastatic breast cancer patients in less than 28 days from consent by evaluating the time to analysis and suggestions
Time to report molecular profiling in blood | 28 days
  2.1.2 To demonstrate the feasibility of real-time molecular profiling of blood samples in metastatic breast cancer patients within 4 weeks from consent to analysis

SECONDARY OUTCOMES:
Ability to make treatment suggestions | 28 days
  To demonstrate the ability to make treatment suggestions based on the molecular profile of patients' tumors
Decisions about Molecular Profiling Tumor Board (MPTB) suggestion | 1 year
  To analyze why clinicians/patients do or do not proceed with the suggestion of the MPTB
Progression-free survival | 1 year
  To describe progression-free survival (PFS) for women who act on the suggestion of the MPTB and for those choosing a different therapy from our suggestion
Changes in plasma tumor DNA (ptDNA) | 1 year
  To prospectively follow plasma tumor DNA in all patients who take part
Similarities and differences of the profiling results with the different assays in tissue | 1 year
  To examine the correlation of a smaller targeted gene panel between Foundation Medicine's assay and Johns Hopkins Molecular Diagnostics Lab assay

OTHER OUTCOMES:
Similarities and differences of the profiling assay results between blood and tissue samples | 1 year
  To examine the concordance of molecular profiling in blood and tissue with Foundation Medicine's assay in patients with previously tested tumor tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States